CLINICAL TRIAL: NCT00565344
Title: Medicaid Disenrollment: Intrastate Emergency Department Impact
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Ben Heavrin, Assistant Professor of Emergency Medicine, Vanderbilt University
Other Study IDs: Medicaid Disenrollment; EMF Resident Research Grant
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2007-11

CONDITIONS: Medicaid Enrollment Status
Keywords: Medicaid; Disenrollment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We will obtain data from the robust Agency for Healthcare Reimbursement and Quality (AHRQ) Healthcare Utilization Project (HCUP), as well as from the State of Tennessee. If our hypotheses are true, such data will provide strong evidence that Medicaid disenrollment has a negetive health impact on uninsured populations. The data may also provide evidence for increased public funding of safety-net EDs after Medicaid disenrollment.

ELIGIBILITY:
Inclusion Criteria:

* data will be obtained from the Agency for Healthcare Reimbursement and Quality (AHRQ) Healthcare Utilization Project (HCUP)

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be obtained through two datbases. All patients visiting an ED in Tennessee over a 3 year period are included.
Sampling Method: Non-Probability Sample
Enrollment: 5000000 (Actual)
Dates: Start 2007-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The proportion of ED visits from uninsured and TennCare patients after TennCare disenrollment | Upon record review
  The proportion of ED visits from uninsured and TennCare patients after TennCare disenrollment

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Heavrin, MD, Principal Investigator — Vanderbilt University Medical Center